CLINICAL TRIAL: NCT05303441
Title: The Predictive and Diagnostic Value of Using Cystatin C and High Sensitive Troponin Level Together for Diagnosis of ACS in Patients With Chronic Kidney Disease Coming to Emergency Department With Chest Pain
Brief Title: The Predictive and Diagnostic Value of Cystatin C and High Sensitive Troponin
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ankara Diskapi Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Bedriye Muge Sonmez, associate professor, Ankara Diskapi Training and Research Hospital
Other Study IDs: AnkaraDiskapiTRH
Record Dates: First submitted 2022-03-09; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Acute Coronary Syndrome; Chronic Kidney Diseases
MeSH Terms: conditions — Acute Coronary Syndrome; Renal Insufficiency, Chronic | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- patients with acute coronary syndrome: patients with chronic kidney disease having chest pain with ecg, symptom or cardiac troponin levels compatible with ACS
  Interventions: Procedure: percutaneous coronary intervention
- patients without acute coronary syndrome: patients with chronic kidney disease having chest pain with ecg, symptom or cardiac troponin levels NONcompatible with ACS

INTERVENTIONS:
Procedure: percutaneous coronary intervention — conventional coronary angiography
  Groups: patients with acute coronary syndrome

SUMMARY:
Our study is planning to evaluate patients with chronic kidney disease who come to the emergency department with chest pain. Estimated GFR (cisGFR) with cystatin and estimated GFR (creaGFR) with creatinine will be calculated. Symptoms, ECG and troponin values of patients will be evaluated for diagnosis of acute coronary syndrome

DETAILED DESCRIPTION:
Our study is planning to evaluate patients with chronic kidney disease who come to the emergency department with chest pain. Estimated GFR (cisGFR) with cystatin and estimated GFR (creaGFR) with creatinine will be calculated. Symptoms, ECG and troponin values of patients will be evaluated for diagnosis of acute coronary syndrome and the final diagnosis of AMI will be adjudicated by 2 independent cardiologists.Serial troponin measurements and eGFR values will be proportioned. These values the will be evaluated and compared for patients with acute coronary syndrome(culprit lesion on conventional coronary angiography) and non-ACS ones . With these data we aim to facilitate the diagnosis of acute coronary syndrome,increase the specificity and sensitivity of cardiac troponins for the diagnosis of acute coronary syndrome of patients with chronic kidney disease, increase the utility of high sensitive troponins for patients with chronic kidney disease. Again, with these data, it is aimed to reduce the number of false negative and false positive diagnosis of acute coronary syndrome .

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18,
2. chronic kidney diease having chest pain or equivalent of chest pain (dyspnea, diaphoresis, syncope, nausea, vomiting) -

Exclusion Criteria:

1. STEMI,
2. age less than 18,
3. missing data,
4. patients referred to or accepted from another medical facility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with chronic kidney disease having chest pain and administered to emergency department for differential diagnosis of chest pain or equivalent of chest pain (dyspnea, diaphoresis, syncope, nausea, vomiting)
Sampling Method: Probability Sample
Enrollment: 172 (Estimated)
Dates: Start 2022-03-07 (Actual); Primary Completion 2023-01-07 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
anticipated ACS | time passed until PCI (percutaneous coronary intervention) (pre-intervention) or admission to hospital
  The role of cystatin C in diagnosis acute coronary syndrome when used with troponin in patients with chronic renal failure.
exclusion of acs | time passed during emergency department visit until discharge avarage of 3-6 hours
  exclusion of ACS according to current guidelines

CONTACTS AND LOCATIONS:
Overall Officials: bedriye müge sönmez, assoc. prof., Study Director — research
Locations (1):
- Diskapi Research and Training Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Hamzacebioglu E, Sonmez BM, Akcay G, Tulmac M, Kayisoglu S, Hatil SI, Gungor EB. Valency of cystatin C and creatinine on troponin values in chronic kidney disease patients with chest pain in emergency department. Am J Emerg Med. 2025 Mar;89:95-102. doi: 10.1016/j.ajem.2024.12.020. Epub 2024 Dec 13. PMID 39705855